CLINICAL TRIAL: NCT05262998
Title: Intramedullary Screw Fixation Versus Plate in Completely Displaced Midshaft Clavicle Fractures ?
Brief Title: Intramedullary Screw Versus Plate in Displaced Midshaft Clavicle Fractures
Acronym: PlaClaVis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bichat Hospital (Other)
Responsible Party: Principal Investigator, Jules Descamps, Medical Doctor, Bichat Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0901-01
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-03

CONDITIONS: Clavicle Fracture
Keywords: Clavicle; Fracture; Screw; Intramedullary; Plate; Trauma; Upper limb
MeSH Terms: conditions — Fractures, Bone; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Active Comparator): Plate fixation
  Interventions: Procedure: Plate fixation
- INTERVENTION (Experimental): Intramedullary Screw
  Interventions: Procedure: Intramedullary Screw

INTERVENTIONS:
Procedure: Plate fixation — Procedure: plate fixation
  Plate fixation was performed by the regular on-call team surgeons and adhered to standard principles of fracture fixation. A standard surgical protocol was used, the approach was moved inferiorly, the fracture was reduced, sometimes with osteosutur and fixed with an antero-superior anatomical plate. 3.5mm Locked and cortical screws were used on both sides of the fracture. Fluoroscopy was used during the procedure. Intradermal suture was used to close the skin
  Other: post-intervention All patients were discharged the day after the surgery. Interruption of work was given for 45 days. The same analgesics were administered in both groups for three weeks. Graduated exercises for the shoulder joint with pendular movements in a range of 15°-20° with the protection of a forearm sling were commenced from the postoperative second day. The sling was removed when X-ray films showed growth of callus or an indistinct fracture line.
  Arms: CONTROL
Procedure: Intramedullary Screw — Procedure: Intramedullary screw fixation
  Intramedullary screw fixation was performed by the regular on-call team surgeons and adhered to standard principles of fracture fixation. Intramedullary screw fixation was performed by using a 1.6 or 2.8 mm-diameter threaded guide pin and a 85-100 mm long, 4.5 or 6.5 mm-diameter cannulated screw tapped in along the guide pin. Fluoroscopy was used during the procedure. Intradermal suture was used to close the skin.
  Other: post-intervention All patients were discharged the day after the surgery. Interruption of work was given for 45 days. The same analgesics were administered in both groups for three weeks. Graduated exercises for the shoulder joint with pendular movements in a range of 15°-20° with the protection of a forearm sling were commenced from the postoperative second day. The sling was removed when X-ray films showed growth of callus or an indistinct fracture line.
  Arms: INTERVENTION

SUMMARY:
This study compares two operative managements of midshaft clavicle fractures: intramedullary screw and plate fixation.

In the past ten years, many studies have compared non operative management versus operative fixation and in particular plate fixation which has been well evaluated. But to date, there are only few retrospective studies that compares plate and intramedullary screw fixation and the knowledge about this last technique and its functional results is poor.

The main objective of this study is to compare plate and intramedullary screw fixation, in term of functional results and rate of union.

The hypothesis of this study is that there is superiority of plate over intramedullary screw fixation.

The main evaluation criterion is the Constant Score at 3 months postoperatively.

DETAILED DESCRIPTION:
Clavicle fractures are common, accounting for about 4% of all fractures, of which 80% occur in the middle third of the bone and occur typically in younger patients, posing a burden for this active population. Traditionally, non-operative treatment with a sling was standard care, however, increasing rates of fixation are now being reported.

Currently, the main procedure for surgical treatment of clavicular fractures is internal fixation with a plate. Plates provide reliable and secure fixation, but require a long incision and usually have to be removed in a second operation. In a meta-analysis of controlled randomized trials conducted by Woltz, the overall rate of secondary intervention in the plate fixation group was elevated at 17.6%, of which 58.9% was for implant removal.

Fuglesang assessed in a randomized controlled trial the functional results of plate fixation versus intramedullary nailing of displaced midshaft clavicle fractures and found that there was no significant difference between the two treatments courses at twelve months and QuickDASH and Constant Score were both excellent in the two groups. They noticed that recovery was faster with plate fixation (QuickDASH significantly better and clinically relevant (inferior by 8.7 points) at 5 weeks of follow-up and QuickDASH and Constant Score significantly better between 6 weeks and 6 months of follow-up).

They highlighted a significant higher rate of complications when a 2mm diameter nail was used for patients with peropertively discovery of narrow medullary canal. Thus, they suggested a conversion to open reduction and internal fixation with a plate when a 2.5 mm nail may not be used. Morever, they showed that degree of comminution was a strong predictor factor of functional results. The more comminution, the higher were the Quick-DASH and DASH scores during the first six months in the intramedullary nailing group. Plating appeared to be able to negate the effect of comminution when bridging the fracture and concluded that in the presence of comminution, plating may be the superior option.

Sun conducted a retrospective study comparing minimally invasive intramedullary fixation with cannulated screws versus plate fixation and showed that time to union was significantly lower in cannulated screw group (13.2 ± 6.9 weeks versus 16.3 ± 8.7 weeks in the plate fixation group) but there was no subsequent significant difference in Neer shoulder activity score between the two groups. Thus, the clinically significance is yet to be assessed.

In the light of the above considerations, we compared the functional results of cannulated screw fixation versus reconstruction plate fixation using a randomized prospective study design.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 yrs
* Midshaft Clavicle fracture
* Completely displaced (one of the criteria)

  * Displacement by one bone width
  * Angulation exceeding 30°
  * Initial shortening of more than 20 mm
  * Tenting/compromised skin

Exclusion Criteria:

* Open fracture of the clavicle
* Fracture > 3 wks old
* Noncompliance
* Substance abuse
* Not a resident in the area surrounding the hospital
* Pathological fracture
* Congenital abnormality/bone disease
* Infectious process around the clavicle area
* Neurovascular injury

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
The Constant Score | At 3 months
  Scale from 0 to 100 to evaluate the shoulder function in daily life (0 is no function and 100 is normal function)

SECONDARY OUTCOMES:
The Constant Score | At 6 weeks, 4 months, 6 months and 12 months
  Scale from 0 to 100 to evaluate the shoulder function in daily life (0 is no function and 100 is normal function)
The QuickDASH Score | At 6 weeks, 3, 4, 6 and 12 months
  Scale from 0 to 100 to evaluate the shoulder function in daily life (0 is no disability and 100 is maximum disability)
Numeric Rating Scale (NRS) | At 6 weeks, 3, 4, 6 and 12 months
  Scale from 0 to 10 to evaluate pain (0 is no pain and 10 is worst pain)
Subjective Shoulder Value | At 6 weeks, 3, 4, 6 and 12 months
  Scale from 0 to 100% to evaluate subjective shoulder assessment (0% is no shoulder function and 100% is normal shoulder)
Time to fracture union | At 6 weeks, 3, 4, 6 and 12 months
  From surgery to union (in days)
Length of incision | Peroperatively
  All incision in cm
The duration of surgery | Peroperatively
  From incision to closure (in min)
Blood loss during surgery | Peroperatively
  Estimation in mL
Cosmetic result, Numeric Rating Scale | At 12 months
  Scale from 0 to 10 to evaluate cosmetic (0 is worst result and 10 perfect result)
Rated satisfaction | At 6 weeks, 3, 4, 6 and 12 months
  1: Very Satisfied ; 2: Satisfied ; 3: Ok ; 4: Dissatisfied ; 5: Very dissatisfied
Rate of secondary surgery or complication for non union, mal union, infection of the operative site and implant removal | At 12 months
  Descriptive

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Boyer, PhD, Study Chair — Bichat Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sun JZ, Zheng GH, Zhao KY. Minimally invasive treatment of clavicular fractures with cannulated screw. Orthop Surg. 2014 May;6(2):121-7. doi: 10.1111/os.12108. PMID 24890294
- [Result] Fuglesang HFS, Flugsrud GB, Randsborg PH, Oord P, Benth JS, Utvag SE. Plate fixation versus intramedullary nailing of completely displaced midshaft fractures of the clavicle: a prospective randomised controlled trial. Bone Joint J. 2017 Aug;99-B(8):1095-1101. doi: 10.1302/0301-620X.99B8.BJJ-2016-1318.R1. PMID 28768788
- [Result] Khalil A. Intramedullary screw fixation for midshaft fractures of the clavicle. Int Orthop. 2009 Oct;33(5):1421-4. doi: 10.1007/s00264-009-0724-2. Epub 2009 Feb 19. PMID 19225778
- [Result] Smith SD, Wijdicks CA, Jansson KS, Boykin RE, Martetschlaeger F, de Meijer PP, Millett PJ, Hackett TR. Stability of mid-shaft clavicle fractures after plate fixation versus intramedullary repair and after hardware removal. Knee Surg Sports Traumatol Arthrosc. 2014 Feb;22(2):448-55. doi: 10.1007/s00167-013-2411-5. Epub 2013 Jan 31. PMID 23370985
- [Result] Domos P, Tytherleigh-Strong G, Van Rensburg L. Increased wound complication with intramedullary screw fixation of clavicle fractures: Is it thermal necrosis? J Orthop Surg (Hong Kong). 2017 Sep-Dec;25(3):2309499017739482. doi: 10.1177/2309499017739482. PMID 29129131